CLINICAL TRIAL: NCT03956914
Title: A 8-weeks, Randomized, Double-blind, Placebo-Controlled, Cross-Over Clinical Trials to Evaluated the Efficacy and Safety of Deep Sea Water on Blood Glucose Level
Brief Title: Efficacy and Safety of Deep Sea Water on the Blood Glucose Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CTCF2_2016_DSW
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSW (deep sea water) group (Experimental): DSW, 440 ml/day for 8 weeks
  Interventions: Other: Deep sea water
- Placebo group (Placebo Comparator): Placebo, 440 ml/day for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placeob water 440 ml/day for 8 weeks
  Arms: Placebo group
Other: Deep sea water — Deep sea water 440 ml/day for 8 weeks
  Arms: DSW (deep sea water) group

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of deep sea water on improvement of hyperglycemia

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled, cross-over clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose concentration of 100-140 mg/dL or 2h-postprandial plasma glucose concentration of 140 ~199 mg/dL

Exclusion Criteria:

* Patients with type 1 or type 2 diabetes
* HbA1c ≥9.0%
* Weight decreased by more than 10% within past 3 months
* Have clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, hepatic biliary system, kidney and Urinary system, neuropsychiatry, musculoskeletal, inflammatory and hematologic malignancies, gastrointestinal disorders, etc.
* Hypoglycemic agent, obesity medicine, lipid lowering agent within past 6 months or functional food within past 2 month
* Subjects who have taken corticosteroid within past 1 months
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test by show the following results

  * Serum AST (aspartate aminotransferase) or ALT (alanine aminotransferase) > 2 times the upper limit of normal range
  * Serum Creatinine > 2.0 mg/dl
* Pregnancy or breast feeding
* If a woman of childbearing doesn't accept the implementation of appropriate contraception
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Changes of blood glucose | Baseline, 8 weeks
  Concentration of fasting and postprandial glucose during OGTT (oral glucose tolerance test) were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of blood insulin | Baseline, 8 weeks
  Concentration of blood insulin were assessed before and after the intervention
C-pepetide | Baseline, 8 weeks
  Concentration of C-peptide were assessed before and after the intervention
HbA1c | Baseline, 8 weeks
  Concentration of HbA1c were assessed before and after the intervention
Homeostatic model assessment - insulin resistance (HOMA-IR) | Baseline, 8 weeks
  Concentration of HOMA-IR were assessed before and after the intervention
Total cholesterol | Baseline, 8 weeks
  Concentration of total cholesterol were assessed before and after the intervention
Triglyceride | Baseline, 8 weeks
  Concentration of triglyceride were assessed before and after the intervention
HDL-cholesterol | Baseline, 8 weeks
  Concentration of HDL-cholesterol were assessed befor and after the intervention
LDL-cholesterol | Baseline, 8 weeks
  Concentration of LDL-cholesterol were assessed befor and after the intervention
Weight | Baseline, 8 weeks
  Concentration of weight were assessed befor and after the intervention
BMI | Baseline, 8 weeks
  Concentration of BMI were assessed before and after the invervention
Body fat mass | Baseline, 8 weeks
  Concentration of body fat mass were assessed before and after the intervention
Percent of body fat mass | Baseline, 8 weeks
  Concentration of percent of body fass mass were assessed before and after the intervention
Waist circumference | Baseline, 8 weeks
  Concentration of waist circumference were assessed before and after the intervention
Waist-hip ratio (WHR) | Baseline, 8 weeks
  Concentration of WHR were assessed before and after the intervention

IPD SHARING:
Plan to Share IPD: No